CLINICAL TRIAL: NCT06696781
Title: NOL Index in Response to Pacemaker Stimulation in Open-heart Surgery
Brief Title: NOL Index in Response to Pacemaker Stimulation
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 33964
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Nociceptive Pain
Keywords: cardiac surgery; nociception; NOL index; pacemaker
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pacemaker: Mechanically ventilated postoperative adult patients, admitted to the intensive care unit (ICU) within 6 hours after elective cardiac surgery, undergo pacemaker stimulation at various rates to observe how this influences the NOL Index.
  Interventions: Procedure: Pacemaker stimulation

INTERVENTIONS:
Procedure: Pacemaker stimulation — We deactivate the pacemaker to establish baseline measurements of NOL, bispectral index (BIS), mean arterial pressure (MAP), and heart rate (HR), recorded every minute for 5 minutes. We then adjust the pacemaker to 90 bpm and 110 bpm in subsequent 5-minute phases to assess the physiological responses. After deactivating the pacemaker to analyze washout effects, we reactivate it at 110 bpm to observe any changes. A temporary disconnection of the NOL monitor for 1 minute tests system reliability, followed by continued monitoring at the same rate for an additional 5 minutes. Each measurement phase averages data from the last 10 seconds each minute to ensure accuracy and reduce artifacts.

SUMMARY:
The Nociception Level Index (NOL Index) utilizes various signals to assess the balance of nociception and antinociception during anesthesia. Its correlation with nociceptive stimuli and opioids is known, but its response to isolated heart rate changes remains uncertain. The aim is to investigate how cardiac pacing affects the NOL Index.

DETAILED DESCRIPTION:
The Nociception Level Index (NOL Index) represents an innovative approach to monitoring nociception during general anesthesia, utilizing a combination of signals from photoplethysmography, accelerometry, thermometry, and skin conductance to assess the balance between nociceptive and antinociceptive states. Research has already established how the NOL Index correlates with both nociceptive stimuli and opioid levels, providing valuable insights into patient responses. However, the impact of changes in heart rate, specifically through isolated cardiac pacing, on the NOL Index is not yet clear. The primary goal of this study is to explore and understand how cardiac pacing might influence the readings of the NOL Index, potentially offering a new dimension to managing anesthesia effectively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Preoperative and postoperative sinus rhythm (50-90 bpm)
* Norepinephrine support < 100 ng/kg/min

Exclusion Criteria:

* Redo or emergent surgery
* History of any cardiac arrhythmia
* Any cardiocirculatory support other than norepinephrine
* Perioperative treatment with beta-blockers, calcium-channel blockers or ivabradine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated postoperative adult patients, admitted to the ICU within 6 hours after elective cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
NOL index | Every minute during seven 5-minute intervals under various pacemaker settings, totaling 35 minutes of monitoring.
  The Nociception Level Index (NOL Index) quantitatively evaluates the balance between nociception and antinociception in mechanically ventilated postoperative adult patients after elective cardiac surgery, utilizing a multiparametric approach that includes photoplethysmography, accelerometry, thermometry, and skin conductance.

CONTACTS AND LOCATIONS:
Overall Officials: Serban-Ion Bubenek-Turconi, Professor, Study Chair — CC Iliescu Cardiovascular Institute
Locations (1):
- "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balan C, Barbulescu RT, Dumitrache A, Fodoroiu A, Morosanu B, Nica A, Stanculea I, Stoian I, Valeanu L, Wong A, Bubenek-Turconi SI. Nociception level index response to pacemaker stimulation. J Clin Monit Comput. 2025 Dec;39(6):1309-1316. doi: 10.1007/s10877-025-01377-w. Epub 2025 Nov 3. PMID 41182599